CLINICAL TRIAL: NCT03292172
Title: Open Label, Dose Finding and Expansion Phase IB Study to Evaluate the Safety, Pharmacokinetics and Clinical Activity of RO6870810 and Atezolizumab (Pd L1 Antibody) in Pateints With Advanced Ovarian Cancer or Triple Negative Breast Cancer
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics and Clinical Activity of RO6870810 and Atezolizumab (PD-L1 Antibody) in Participants With Advanced Ovarian Cancer or Triple Negative Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Portfolio prioritization
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NP39487; 2017-001147-13 (EudraCT Number)
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Advanced Ovarian Cancer; Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — atezolizumab; RO6870810

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 - Escalation Dose: RO6870810 + Atezolizumab (Experimental): Participants will be administered escalating doses of RO6870810 (0.3 milligram per kilogram [mg/kg], 0.45 mg/kg, and 0.65 mg/kg) subcutaneously (SC) once daily (QD) along with fixed dose of atezolizumab 1200 mg intravenously (IV) on Day 1 of each cycle (21 day cycles), every 3 weeks. RO6870810 will be given during the first 14 days.
  Interventions: Drug: Atezolizumab; Drug: RO6870810
- Group 2 - Sequential Dose: RO6870810 + Atezolizumab (Experimental): Participants will be administered RO6870810 monotherapy (starting dose 0.30 mg/kg) during the first 14 days of 21-day Run-in period. Following the Run-in period, participants will continue to receive RO6870810 at the same dose in combination with fixed dose of atezolizumab 1200 mg IV every 3 weeks in 21-day cycles.
  Interventions: Drug: Atezolizumab; Drug: RO6870810
- Group 3 - Expansion in TNBC Group: RO6870810 + Atezolizumab (Experimental): Participants will be administered dose of RO6870810 established in Group 1 (either 0.3 mg/kg, 0.45 mg/kg, or 0.65 mg/kg) SC QD along with fixed dose of atezolizumab 1200 mg IV on Day 1 of each cycle (21 day cycles), every 3 weeks. RO6870810 will be given during the first 14 days.
  Interventions: Drug: Atezolizumab; Drug: RO6870810
- Group 4 - Expansion in OC Group: RO6870810 + Atezolizumab (Experimental): Participants will be administered dose of RO6870810 established in Group 1 (either 0.3 mg/kg, 0.45 mg/kg, or 0.65 mg/kg) SC QD along with fixed dose of atezolizumab 1200 mg IV on Day 1 of each cycle (21 day cycles), every 3 weeks. RO6870810 will be given during the first 14 days.
  Interventions: Drug: Atezolizumab; Drug: RO6870810

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be given intravenously (IV) at a fixed dose of 1200 mg on Day 1 of each cycle, every 3 weeks.
Drug: RO6870810 — RO6870810 will be injected SC,at initial planned doses of 0.30, 0.45, or 0.65 mg/kg, QD for the first 14 days of a 21-day cycle.

SUMMARY:
This is Phase IB, open label, non-randomized study designed to investigate the dose, safety, pharmacokinetics and anti-tumor activity of RO6870810 in combination with a fixed dose of atezolizumab. The study consists of four groups, Group 1 (Dose Escalation Group) and Group 2 (Sequential Dose Group), and Groups 3 and 4 (Expansion Groups), which will further evaluate the safety, pharmacokinetic, pharmacodynamic and preliminary clinical activity in patients with triple negaive breast cancer and/or ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:-

* Groups 1 and 2: Participants with histologically confirmed advanced ovarian cancer or triple negative breast cancer who in the opinion of the Investigator are appropriate for this study
* Group 3: Participants with histologically confirmed TNBC who have received either one or 2 prior systemic treatments for metastatic breast cancer, and who have documented disease progression on or after the most recent treatment
* Group 4: Recurrent ovarian cancer participant who have received no more than two prior lines of platinum therapy in the recurrent setting and have progressed within 9 months from the last platinum containing regimen
* Measurable disease by RECIST criteria version 1.1 prior to study drug administration
* Performance status of 0 or 1 on the eastern Cooperative Oncology Group (ECOG) scale
* Life expectancy, in the opinion of the Investigator, of at least 3 months
* Disease-free of active second/secondary or prior malignancies for => 2 years with the exception of squamous cell carcinoma of the skin, or carcinoma in situ of the cervix or breast
* Willing to provide the protocol specified tumor biopsies
* Acceptable hematologic status, liver and renal function
* Groups 1 and 2: Participants who have received prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies, may be enrolled, provided the following requirements are met:

  * Minimum of 5 months from the last dose of anti-PD-1, anti-CTLA-4, anti-PD- L1 or CD137 agonist treatment
  * No history of severe immune-related adverse effects from CD137 agonist, anti-CTLA-4, anti-PD-1 or anti-PD-L1 (NCI CTCAE Grade 3 and 4). Any toxicity related to the therapy must have resolved completely, no residual toxicity as assessed by NCI CTCAE (v4.03)
* Agree to use protocol defined methods of contraception - For all participants, the reliability of sexual abstinence must be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the participant. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not acceptable methods of contraception

Exclusion Criteria:

* Participants with history of prior malignancy except solid tumor treated curatively more than 3 years ago without evidence of recurrence
* Asymptomatic or symptomatic, untreated, or actively progressing central nervous system (CNS) metastases
* History of leptomeningeal disease
* Uncontrolled tumor-related pain
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures. Participants with indwelling catheters are allowed.
* Uncontrolled or symptomatic hypercalcemia
* New York Heart Association Class III or IV cardiac disease, pericarditis, myocardial infarction within the past 6 months, unstable arrhythmia
* Fredericia-corrected QT interval (QTcF) > 470 milli seconds (msec) (female) or > 450 msec (male), or history of congenital long QT syndrome. Any electrocardiogram (ECG) abnormality, including pericarditis, which in the opinion of the Investigator would preclude safe participation in the study.
* Active, uncontrolled bacterial, viral, or fungal infections within 7 days of study entry requiring systemic therapy. Participants with active TB infection are excluded from the study.
* Known clinically important respiratory impairment
* History of major organ transplant
* History of an autologous or allogeneic bone marrow transplant
* Serious non-malignant disease that could compromise protocol objectives in the opinion of the Investigator and/or the Sponsor
* Pregnant or nursing women
* Any systemic anticancer therapy within 3 weeks prior to Cycle 1 Day 1
* Any radiation treatment to metastatic site within <= 14 days of Cycle 1 Day 1
* Major surgical procedure, open biopsy, or significant traumatic injury within 30 days prior to Cycle 1 Day 1 or anticipation of need for major surgical procedure during the course of the study
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric, human or humanized antibodies or fusion proteins
* Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation
* Active or history of autoimmune disease
* History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest computed tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Positive test for Human immunodeficiency virus (HIV)
* Active hepatitis B or hepatitis C
* Receipt of a live, attenuated vaccine within 4 weeks prior to randomization or anticipation that such a live, attenuated vaccine will be required during the study
* Treatment with investigational therapy within 28 days prior to initiation of study treatment
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment
* Consumption of agents which strongly inhibit CYP3A4 enzyme, within 7 days prior to the first dose of study treatment and during the study
* Consumption of agents which strongly induce CYP3A4 enzyme, within 14 days prior to the first dose of study treatment and during the study
* Treatment with systemic immuno-stimulatory agents within 4 weeks or five half-lives of the drug (whichever is shorter) prior to the first dose of study treatment
* Treatment with systemic corticosteroids or other systemic immunosuppressive medications within 2 weeks prior to the first dose of study treatment, or, anticipated requirement for systemic immunosuppressive medications during the trial
* History of allergic reactions attributed to components of the formulated product(s)
* Unwillingness or inability to comply with procedures required in this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2019-02-26 (Actual); Study Completion 2019-02-26 (Actual)

PRIMARY OUTCOMES:
Group 1: Percentage of Participants With Dose Limiting Toxicities (DLT) | Cycle 1 (Day 21)
Groups 1 to 4: Percentage of Participants With Adverse Events (AEs) | Up to 22 months
Groups 1 to 4: Percentage of Participants With Change in Vital Signs, Physical Findings, Electrocardiogram (ECG) and Laboratory Parameters | Baseline up to follow-up visit (approximately 22 months)
Groups 3 and 4: Objective Response (OR) as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. | From first occurrence of objective response until disease progression or death from any cause (Up to 22 months)

SECONDARY OUTCOMES:
Groups 1 to 4: Maximum concentration (Cmax) of RO6870810 (RO) and Atezolizumab (Ate) | RO: Pre-dose Day 1,14,21;0.25,0.5,1,2,4,6,8,10hour (h) post-dose Day 14;24,28h post-dose Day 15 Run-in, Cycle 1, even cycles till end of treatment; Ate: pre-dose, end of infusion Day 1 Cycle 1; pre-dose Day 1 of even cycles; follow-up (Up to 22 months)
Groups 1 to 4: Time of maximum concentration (tmax) of RO6870810 and Atezolizumab | RO: Pre-dose Day 1,14,21;0.25,0.5,1,2,4,6,8,10hour (h) post-dose Day 14;24,28h post-dose Day 15 Run-in, Cycle 1, even cycles till end of treatment; Ate: pre-dose, end of infusion Day 1 Cycle 1; pre-dose Day 1 of even cycles; follow-up (Up to 22 months)
Groups 1 to 4: Clearance (CL) or Apparent Clearance (CL/F) of RO6870810 and Atezolizumab | RO: Pre-dose Day 1,14,21;0.25,0.5,1,2,4,6,8,10hour (h) post-dose Day 14;24,28h post-dose Day 15 Run-in, Cycle 1, even cycles till end of treatment; Ate: pre-dose, end of infusion Day 1 Cycle 1; pre-dose Day 1 of even cycles; follow-up (Up to 22 months)
Groups 1 to 4: Volume of Distribution (Vd) or Apparent Volume of Distribution (Vd/F) of RO6870810 and Atezolizumab | RO: Pre-dose Day 1,14,21;0.25,0.5,1,2,4,6,8,10hour (h) post-dose Day 14;24,28h post-dose Day 15 Run-in, Cycle 1, even cycles till end of treatment; Ate: pre-dose, end of infusion Day 1 Cycle 1; pre-dose Day 1 of even cycles; follow-up (Up to 22 months)
Groups 1 to 4: Area Under the Plasma Concentration-Time Curve From Time Zero to End of the Dosing Interval (AUC0-tau) of RO6870810 and Atezolizumab | RO: Pre-dose Day 1,14,21;0.25,0.5,1,2,4,6,8,10hour (h) post-dose Day 14;24,28h post-dose Day 15 Run-in, Cycle 1, even cycles till end of treatment; Ate: pre-dose, end of infusion Day 1 Cycle 1; pre-dose Day 1 of even cycles; follow-up (Up to 22 months)
Groups 1 to 4: Area Under the Plasma Concentration Time Curve From Time Zero to Infinity (AUC0-inf) of RO6870810 and Atezolizumab | RO: Pre-dose Day 1,14,21;0.25,0.5,1,2,4,6,8,10hour (h) post-dose Day 14;24,28h post-dose Day 15 Run-in, Cycle 1, even cycles till end of treatment; Ate: pre-dose, end of infusion Day 1 Cycle 1; pre-dose Day 1 of even cycles; follow-up (Up to 22 months)
Groups 1 to 4: Half life (t1/2) of RO6870810 and Atezolizumab | RO: Pre-dose Day 1,14,21;0.25,0.5,1,2,4,6,8,10hour (h) post-dose Day 14;24,28h post-dose Day 15 Run-in, Cycle 1, even cycles till end of treatment; Ate: pre-dose, end of infusion Day 1 Cycle 1; pre-dose Day 1 of even cycles; follow-up (Up to 22 months)
Groups 1 to 4: Trough concentration (Ctrough) of RO6870810 and Atezolizumab | Pre-dose at Cycle 2 and at the beginning of every subsequent even-number cycles (Up to 22 months)
Groups 1 and 2: Objective Response (OR) as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. | From first occurrence of objective response until disease progression or death from any cause (Up to 22 months)
Groups 1 to 4: Objective Response (OR) as per Immune-Modified RECIST | From first occurrence of objective response until disease progression or death from any cause (Up to 22 months)
Groups 1 to 4: Duration of Response (DoR) as per RECIST v1.1 and Immune-Modified RECIST | From first occurrence of objective response until disease progression or death from any cause (Up to 22 months)
Groups 1 to 4: Progression-Free Survival (PFS) per RECIST v1.1 and Immune-Modified RECIST | From first occurrence of objective response until disease progression or death from any cause (Up to 22 months)
Groups 1 to 4: Overall Survival (OS) | From the time of first dose of study treatment to the time of death from any cause (Up to 22 months)
Groups 1 to 4: Tumor Marker Assessments (CA-125, According to Modified Gynecologic Cancer InterGroup [GCIG] Guidelines,CEA, CA15-3 Changes) | Day 1 of each cycle till end of treatment or disease progression or death from any cause (Up to 22 months)
Groups 1 to 4: Changes in CD11b Expression Levels Measurement in CD14+ Monocytes From Blood Association with Steady-State RO6870810 PK Drug Exposure | Day 1, 8, 15, 21 of Run-in period , Cycle 1
Groups 1 to 4: Changes in Markers (e.g., PD-L1, CD8/Ki 67) in Tissue Biopsy Specimens by Immunohistochemistry (IHC) | Day 1, 15, 21 of Run-in period, Cycle 1
Groups 1 to 4: Percentage of Participants With Transcript Profiling Assessment Receiving Combination Study Treatment | Pre-dose Day 1, 21 Run-in period, Cycle 1; 6h post-dose Day 1 Run-in period, Cycle 1

CONTACTS AND LOCATIONS:
Locations (11):
- United States (3):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Oklahoma University Health Sciences Center, Oklahoma City, Oklahoma
  - Sarah Cannon Res Inst; TN Onc, Nashville, Tennessee
- Australia (2):
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Peter MacCallum Cancer Centre; Medical Oncology, Melbourne, Victoria
- University Health Network; Princess Margaret Hospital; Medical Oncology Dept, Toronto, Ontario, Canada
- Rigshospitalet; Onkologisk Klinik, København Ø, Denmark
- United Kingdom (4):
  - Western General Hospital, Edinburgh
  - Guys and St Thomas NHS Foundation Trust, Guys Hospital, London
  - The Christie, Manchester
  - Churchill Hospital, Oxford

REFERENCES:
- [Derived] Marbach D, Brouer-Visser J, Brennan L, Wilson S, Davydov II, Staedler N, Duarte J, Martinez Quetglas I, Nuesch E, Canamero M, Chesne E, Au-Yeung G, Hamilton E, Lheureux S, Richardson DL, Spanggaard I, Gomes B, Franjkovic I, DeMario M, Kornacker M, Lechner K. Immune modulation in solid tumors: a phase 1b study of RO6870810 (BET inhibitor) and atezolizumab (PD-L1 inhibitor). BMC Cancer. 2025 Mar 18;25(1):500. doi: 10.1186/s12885-025-13851-4. PMID 40102759